CLINICAL TRIAL: NCT00506129
Title: Study of Allogeneic Transplantation in Patients With Cutaneous T-Cell Lymphoma (CTCL)
Brief Title: Allogeneic Transplantation in Patients With Cutaneous T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM03-0279; NCI-2012-01547 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Lymphoma; Disorder Related to Bone Marrow Transplantation
Keywords: Cutaneous T-Cell Lymphoma; CTCL; Allogeneic Transplantation; Lymphoma; Allogeneic peripheral blood progenitor cell; PBPC; Bone Marrow transplantation; Stem Cell Transplant; SCT; Fludarabine; Fludarabine Phosphate; Fludara; Melphalan
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Cutaneous | interventions — fludarabine; fludarabine phosphate; Melphalan; Transplantation, Homologous; Bone Marrow Transplantation; Stem Cell Transplantation; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fludarabine + Melphalan with PBPC (Experimental): Fludarabine 25 mg/m^2 intravenous (IV) daily for 5 Days prior to Allogeneic Transplant, Melphalan 70 mg/m^2 IV daily for 2 Days prior to IV Allogeneic Transplant following Fludarabine & Melphalan. Thymoglobulin 2 mg/kg/day IV on days -3, -2 & -1 for patients receiving matched unrelated marrow/stem cells or mismatched related marrow.
  Interventions: Drug: Fludarabine; Drug: Melphalan; Procedure: Allogeneic Transplant; Drug: Thymoglobulin

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 Given By Vein Daily for 5 Days Prior to Allogeneic Transplant.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Melphalan — 70 mg/m^2 Given By Vein Daily for 2 Days Prior to Allogeneic Transplant.
Procedure: Allogeneic Transplant — Allogeneic transplant given by vein after completion of Fludarabine and Melphalan.
  Other Names: Allogeneic peripheral blood progenitor cell; PBPC; Bone Marrow transplantation; Stem Cell Transplant; SCT
Drug: Thymoglobulin — 2 mg/kg/day by vein on days -3, -2 and -1 for patients receiving matched unrelated marrow/stem cells or mismatched related marrow.
  Other Names: ATG; Antithymocyte Globulin

SUMMARY:
The goal of this clinical research study is to see if receiving a transplant of blood stem cells (cells that can produce blood) or bone marrow from either a related donor (brother, sister or other relative) or an unrelated voluntary donor will help patients with advanced cutaneous T-cell lymphoma. The length of time that patients who receive the treatment remain free of disease will also be studied.

DETAILED DESCRIPTION:
You will receive the chemotherapy drug fludarabine for 5 days (Days 1 to 5). The drug melphalan will be given on Days 4 and 5. You may also receive the drug anti-thymocyte globulin (ATG) on Days 4, 5, 6. This will be followed by infusion of blood stem cells or bone marrow from a donor on Day 7. A separate consent will be provided to the donor. The donor can be a brother, sister or another family member or a compatible unrelated donor. The drugs and the stem cells will be given through a catheter (a small tube) placed under the collarbone. You may receive your treatment on an inpatient or outpatient basis. If treated on an inpatient basis, you will stay in the hospital during treatment and recovery, which can take 4 to 5 weeks even if there are no complications.

The chemotherapy and the ATG are given to help the body accept the transplanted stem cells or bone marrow. You will receive antibiotics to fight infection and a medicine called G-CSF (Neupogen®) to help blood counts rise back to healthier levels. G-CSF is given as an injection under the skin. You will also need blood and platelet transfusions.

You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

If the cancer grows and graft-versus-host disease is not present, you may be eligible to receive donor blood cells (lymphocytes) infused through the catheter. This may cause graft-versus-host disease and may help shrink the cancer. If the cancer grows and graft-versus-host disease is already present, then donor lymphocytes are not given.

Sometimes, the body rejects the donor cells; this reaction is called "graft rejection". Sometimes the donor cells attack the body, a reaction called graft-versus-host disease (GvHD). The drugs tacrolimus and methotrexate will be given to help prevent these reactions from occurring. These drugs are given through a vein or by mouth before and/or after the transplant.

You must stay in the Houston area for at least 100 days after the transplant. After 100 days, you must return to Houston every 3 months for 2 years for tests and checkups, then once a year for at least 3 years. If there is no sign of lymphoma growth at the follow up visit(s), you will receive no further treatment.

This is an investigational study. The drugs used in this study are approved by the FDA and are commercially available. As many as 35 patients will take part in the study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically proven cutaneous T-cell lymphoma (CTCL), disease stage IIB to IVB, patients must be in at least a partial response-PR (skin and lymph nodes) after receiving other non-allogeneic transplant therapy, age </= 70 years, Zubrod performance status 0 or 1, left ventricular ejection fraction >/= 50% or approved for transplant by a cardiologist, DLCO >/= 50% predicted or approved for transplant by a pulmonologist, serum creatinine </= 1.5 mg/dL, serum bilirubin < 2mg/dL. SGPT < 3 x upper limit of normal, and no previous history of allogeneic transplantation.
2. Donor: HLA-compatible related (HLA-A, -B, -DRB1 matched or with one-antigen mismatch) or HLA-compatible unrelated (HLA-A, -B, -C and -DRB1 matched or with one-antigen mismatch).

Exclusion Criteria:

1) Patients cannot have active central nervous system (CNS) disease.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2003-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra M. Hosing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Hosing C, Bassett R, Dabaja B, Talpur R, Alousi A, Ciurea S, Popat U, Qazilbash M, Shpall EJ, Oki Y, Nieto Y, Pinnix C, Fanale M, Maadani F, Donato M, Champlin R, Duvic M. Allogeneic stem-cell transplantation in patients with cutaneous lymphoma: updated results from a single institution. Ann Oncol. 2015 Dec;26(12):2490-5. doi: 10.1093/annonc/mdv473. Epub 2015 Sep 28. PMID 26416896
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 26, 2003 to November 05, 2012. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Fludarabine + Melphalan With PBPC: Fludarabine 25 mg/m^2 intravenous (IV) daily for 5 days prior to allogeneic peripheral blood progenitor cell (PBPC) , Melphalan 70 mg/m^2 IV daily for 2 days prior to IV Allogeneic Transplant following Fludarabine & Melphalan. Thymoglobulin 2 mg/kg/day IV on days -3, -2 & -1 for patients receiving matched unrelated marrow/stem cells or mismatched related marrow.
Period: Overall Study
Arm/Group | Fludarabine + Melphalan With PBPC
Started | 33
Completed | 11
Not Completed | 22
Not completed — Disease Progression/Relapse | 15
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Arm/Group | Fludarabine + Melphalan With PBPC
Number analyzed (Participants) | 33
Age, Continuous [Median (Full Range); unit: years] | 55 [20 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Participant's Response According to Physician's Global Assessment of Clinical Condition (PGA)
Description: Response defined by Physician's Global Assessment of Clinical Condition (PGA) where Complete Response (CR) is No evidence of disease; 100% improvement; Partial Response (PR), one of following: 1) Very significant clearance ( > 90% to < 100%); only traces of disease remains; 2) Significant improvement ( > 75% to < 90%); some evidence of disease remain; 3) Intermediate between slight and marked improvement; ( > 50% to < 75%); 4) Some improvement ( > 25% to < 50%); however, significant evidence of disease remains; Stable Disease (SD): Disease has not changed from baseline condition (+<25%); Progressive Disease (PD): Disease is worse than at baseline evaluation by > 25% or more. Response confirmed by a second assessment at least 4 weeks following it. Assessments at baseline, pre and post transplant (100 days) then till disease progression or year one.
Time Frame: Response assessed pre-transplant and 100 days post transplant with follow up at 1 year.
Measure: Number; unit: participants
Arm/Group | Fludarabine + Melphalan With PBPC
Number analyzed (Participants) | 33
participants
  Complete Response (CR) Converted Post Transplant | 19
  CR Prior to Transplant | 6
  Partial Response (PR) | 0
  Stable Disease (SD) | 0
  Progressive Disease (PD) | 16

2. Secondary Outcome: Average Overall Survival (OS) Length
Description: OS was defined as the time from transplantation to the date of death from any cause or last follow up, measured in days.
Time Frame: Baseline to disease progression, followed up to 5 years post transplant
Population: Baseline to disease progression, followed up to 5 years post transplant (assess at 100 days, every 3 months for 2 years, then once a year for at least 3 years)
Measure: Mean (Full Range); unit: Days
Arm/Group | Fludarabine + Melphalan With PBPC
Number analyzed (Participants) | 33
Days | 1207 [17 to 1825]

ADVERSE EVENTS:
Time Frame: Adverse events collected till 30 days following end of active treatment (the date of the stem cell infusion).
Arm/Group | Fludarabine + Melphalan With PBPC
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 33/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fludarabine + Melphalan With PBPC (N=33)
Primary graft failure with autologous reconstitution (Cardiac disorders) | 1 (1)
Cardiac Edema (Cardiac disorders) | 6 (6)
Cardiac Function (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 7 (7)
Congestive heart failure (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
pericarditis (Cardiac disorders) | 1 (1)
tachycardia (Cardiac disorders) | 2 (2)
fever (General disorders) | 8 (8)
fatigue (General disorders) | 5 (5)
fluid overload: Edema (General disorders) | 10 (10)
rigors (General disorders) | 4 (4)
anorexia (Metabolism and nutrition disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 27 (27)
mucositis (Gastrointestinal disorders) | 18 (18)
flatulence (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 32 (32)
constipation (Gastrointestinal disorders) | 2 (2)
dry mouth (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal disorder, GvHD (Gastrointestinal disorders) | 1 (1)
pain (General disorders) | 5 (5)
vomit (Gastrointestinal disorders) | 5 (5)
bladder (Renal and urinary disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 8 (8)
frequency, urine (Renal and urinary disorders) | 2 (2)
hemorrhagic cystitis (Renal and urinary disorders) | 3 (4)
Acute Kidney Disease (renal disorder), dialysis (Renal and urinary disorders) | 1 (1)
abdomen pain (General disorders) | 1 (1)
dysuria (Renal and urinary disorders) | 1 (1)
transaminitis (Hepatobiliary disorders) | 29 (29) — Elevated transaminases alanine transaminase (ALT) and aspartate transaminase (AST)
increase T bilirubin (Investigations) | 6 (6)
infection (Infections and infestations) | 17 (37)
neutropenic fever (Blood and lymphatic system disorders) | 3 (3)
hyperglycemia (Metabolism and nutrition disorders) | 5 (5)
constipation (Gastrointestinal disorders) | 1 (1)
drowsiness (Nervous system disorders) | 2 (2)
dizziness (Nervous system disorders) | 1 (1)
headache (Nervous system disorders) | 13 (13)
anxiety (Psychiatric disorders) | 2 (2)
weakness, generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
muscular wasting (Musculoskeletal and connective tissue disorders) | 1 (2)
myalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
pain (General disorders) | 3 (4)
bone pain (Musculoskeletal and connective tissue disorders) | 5 (5)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hiccoups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Graft versus Host Disease (Injury, poisoning and procedural complications) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes